CLINICAL TRIAL: NCT07113626
Title: Adapting An Evidence-Based Intervention To Improve HIV Testing And PrEP Uptake In Vietnam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of North Carolina, Chapel Hill (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1521; 1K43TW012850-01 (NIH)
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intervention; Control Condition
Keywords: young men who have sex with men; HIV/AIDS; HIV testing; PrEP; mHealth; Vietnam
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Those assigned to the intervention arm will receive access to the adapted HealthMindr app with key features, including HIV test planning, initial risk/PrEP eligibility assessment, ordering of free condoms and HIV test kits, information about PrEP, PrEP provider and HIV testing locations, and any additional features added through the adaptation process. The staff will help participants download the app and walk them through its use during the study visit. These participants will be encouraged to use the app for a period of 3 months. In addition, participants will be provided standard-of-care HIV prevention information upon enrollment at the study site by a study staff, which includes written prevention materials for HIV testing and referrals to local HIV prevention services. Anyone who seroconverts during the study period will be referred to appropriate HIV treatment services.
  Interventions: Behavioral: Mobile app
- Control (No Intervention): Participants randomized to the control arm will be provided standard-of-care HIV prevention information upon enrollment at the study site by a study staff, which includes written prevention materials for HIV testing and referrals to local HIV prevention services. Anyone who seroconverts during the study period will be referred to appropriate HIV treatment services.

INTERVENTIONS:
Behavioral: Mobile app — The intervention will be a mobile app adapted from HealthMindr - an app based on Social Cognitive Theory - for young men who have sex with men in Vietnam. The app, which was developed and tested in the US, offers a range of testing and prevention services, including self-screening for HIV and sexually transmitted infection (STI) risk, a scheduling and reminder system for HIV/ STI testing, PrEP eligibility screener, an ordering platform for delivery of at-home test kits and condoms, and locators for HIV services. Additional features and contents might be revised and added depending on the needs of young men who have sex with men in Vietnam.
  Arms: Intervention

SUMMARY:
Young men who have sex with men are experiencing an ongoing HIV epidemic in Vietnam, with an HIV prevalence of 12%. However, HIV testing and pre-exposure prophylaxis (PrEP) use among young men who have sex with men remain low. To improve HIV testing and PrEP use, mobile health (mHealth) interventions hold great promise to reach young men who have sex with men in low- and middle-income countries. HealthMindr, an evidence-based mHealth intervention developed in the United States for men who have sex with men, is an ideal option for adaptation for young men who have sex with men in Vietnam. The specific aims are to (1) Adapt the HealthMindr app to improve HIV testing and PrEP uptake among young men who have sex with men in Vietnam; (2) Examine acceptability, feasibility and preliminary effectiveness of the adapted app among young men who have sex with men in Vietnam and (3) Explore barriers and facilitators of implementing the adapted app among young men who have sex with men in Vietnam. In Aim 1, theater testing will be conducted through focus group discussions with young men who have sex with men and key other stakeholders, including health officials, clinic staff and community-based organizations. Theater testing data will be used to refine the app for beta testing. During beta testing, a small group of young men who have sex with men will use the app for 30 days, then complete an online survey and an exit interview to rate the app's usability, provide their perspectives of the app and report any other areas for improvement. App analytics will also be collected to understand whether and how the app is used. In Aim 2, the adapted app with be tested among young men who have sex with men through a randomized controlled design. Young men who have sex with men will be randomized into the intervention or control arm (1:1 ratio). The intervention arm will have full access to the app for 3 months, while the control group will receive standard-of-care HIV services. Key app features include HIV test planning, risk and PrEP eligibility assessment, ordering of free condoms and HIV test kits, information about PrEP, and PrEP provider and HIV testing locations. HIV testing and PrEP use will be assessed at baseline and 3 months and compared between groups. A mixed methods approach will be used to evaluate app acceptability and feasibility. Quantitative data on acceptability and feasibility will be collected through the 3-month online survey, while qualitative data will be collected through in-depth interviews with a subset of young men who have sex with men in the intervention arm and other key stakeholders. In Aim 3, through the same qualitative study as Aim 2, factors that influence the implementation of the app will be explored. Determinants from seven domains will be identified: condition, technology, value proposition, adopter system, health organization, wider system and embedding/adaption over time. Only when mHealth interventions are both effective and adopted can they maximize their potential to reduce HIV incidence among target populations. This proposal will generate data for designing a full-scale hybrid type 1 effectiveness-implementation trial to test the adapted app and identify implementation strategies to address the barriers of app implementation in low and middle-income countries.

ELIGIBILITY:
Inclusion Criteria:

* Young men who have sex with men (YMSM):

Theater testing. YMSM are eligible if they (1) are 18-24 years old Vietnamese male; (2) report having anal intercourse with another man in the last 6 months; (3) are HIV negative or of unknown HIV status; (4) own a smartphone; (5) currently live in Hanoi, (6) are able to read and understand Vietnamese without assistance, and (7) are willing to provide informed consent.

Beta testing. Eligibility is similar to theater testing. Randomized controlled trial (RCT). YMSM are eligible if they (1) are 18-24 years old Vietnamese male; (2) report having anal intercourse with another man in the last 6 months; (3) are HIV negative or of unknown HIV status; (4) own a smartphone; (5) currently live in Hanoi, (6) are able to read and understand Vietnamese without assistance, and (7) are willing to provide informed consent and (8) are not being currently on pre-exposure prophylaxis (PrEP).

* Other key stakeholders:

Eligibility criteria of this group are (1) having worked with MSM-related health issues at an HIV/PrEP clinic or community-based organizations (CBO) for at least 6 months and (2) willingness to provide informed consent.

Exclusion Criteria:

* Young men who have sex with men (YMSM):

Theater testing. None Beta testing. Participants will be deemed ineligible if they are unwilling to provide contact information.

Randomized controlled trial. Exclusion criteria include (1) unwilling to provide contact information; (2) currently enrolled in other HIV testing or PrEP program/intervention.

* Other key stakeholders: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 3 months
  Mean score on the 10-item System Usability Scale (for the app) of participants in the intervention arm. Data from this scale will be scored from 0 to 100, and a score of ≥50 indicates that the app is acceptable (higher score means better outcome).
Feasibility (App usage) | 3 months
  The proportion of participants assigned to the intervention arm who open the app at least once during the follow-up period
HIV testing | Baseline; 3 months
  The proportion of participants who get tested for HIV in the last 3 months
PrEP uptake | 3 months
  The proportion of participants who initiate PrEP during the follow-up period

SECONDARY OUTCOMES:
STI testing | Baseline; 3 months
  The proportion of participants who get tested for STI other than HIV in the last 3 months
PrEP clinic visit | Baseline; 3 months
  Number of visit to a PrEP clinic in the last 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided